CLINICAL TRIAL: NCT03107793
Title: Study of Treat to Target Versus Routine Care Maintenance Strategies in Crohn's Disease Patients Treated With Ustekinumab
Acronym: STARDUST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108276; 2016-002918-43 (EudraCT Number); CNTO1275CRD3005 (Other: Janssen-Cilag Ltd.)
Record Dates: First submitted 2017-03-28; First posted 2017-04-11 (Actual); Results first posted 2021-05-19 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Ustekinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- All Participants (Experimental): At Week (Wk) 0, all eligible participants will initiate intravenous (IV) induction treatment with ustekinumab (UST) on a weight-tiered basis at a dose of approximately 6 milligram per kilogram (mg/kg). At Week 8, all participants will receive a 90 milligram (mg) subcutaneous (SC) injection of ustekinumab. At Week 16, participants who do not achieve a Crohn's Disease Activity Index (CDAI) improvement of greater than or equal to (>=) 70 points versus Week 0 (CDAI 70) will leave the study. Remaining participants will be randomized in a 1:1 ratio to either one of two arms for open label maintenance treatment up to Week 48: the treat to target arm or the routine care arm. From Week 48, participants will continue ustekinumab treatment in the study extension period, up to Week 104. Dosing frequency will be adjusted in the extension period for the participants failing to meet the treatment target.
  Interventions: Drug: Ustekinumab
- Routine Care Arm (Experimental): In the routine care arm, assessment visits will be scheduled according to the timing of maintenance treatment injections up to Week 48, which will be in compliance with the EU SmPC for ustekinumab for the treatment of Crohn's disease, in which dosing every 12 weeks is recommended. At Week 16, (that is, 8 weeks after the first SC dose) participants continuing in the study will have demonstrated a CDAI-70 response. Nonetheless, participants who have not shown adequate response based on the investigator's judgment may receive a second SC dose at Week 16. During the routine care maintenance treatment period, in case of clinical worsening reported by the participant, consistent with disease flare in the investigator's judgment, clinical assessments of disease flare will be performed at the investigator's discretion.
  Interventions: Drug: Ustekinumab
- Treat to Target (T2T) Arm (Experimental): UST maintenance treatment assignment will be based on centrally-read colonoscopy (at Wk16). Participants with <25% improvement in SES-CD score at Wk16 will be assigned to Q8 (8-weekly) treatment and will receive UST 90mg SC at Wk16. In contrast, participants with >=25% improvement in SES-CD score at Wk16 will be assigned to Q12 treatment and will receive next UST dose (90 mg SC) at Wk20. At assessment visits (from Wk24 for participants assigned to the Q8 regimen or from Wk20 for the Q12 group) UST maintenance treatment (up to Wk 48) will be directed by T2T assessments. Participants meeting target will continue with same UST dosing frequency. The dosing frequency will be optimized for all participants failing to meet the target at assessment visit. Those previously on Q12 regimens will be adjusted to Q8 dosing; those previously on Q8 regimens will be adjusted to Q4 dosing. Participants subsequently failing to meet the target will not be able to adjust further and will leave the study.
  Interventions: Drug: Ustekinumab
- Exploratory Extension period: From Week 48 to Week 104 (Experimental): At Week 48, dose de-escalation will be implemented for participants with both endoscopic remission (SES-CD score <=2) and corticosteroid-free clinical remission of at least 16 weeks duration. Participants receiving 12 weekly dosing frequency (Q12) ustekinumab will maintain this dosing frequency. Participants with either clinical remission or endoscopic remission, but not both, at Week 48 will continue with same dosing frequency or de-escalate provided maintenance of corticosteroid-free clinical remission and biomarker remission at 2 consecutive visits. Participants with neither corticosteroid-free clinical remission nor endoscopic remission will escalate dose or leave study if already on 4 weekly dosing frequency (Q4) dose. If neither clinical remission nor biomarker remission is evident at the next visit, participant will leave study. Later in the extension period, only those who achieve corticosteroid-free clinical remission and biomarker remission will undergo dose de-escalation.
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — Participants will receive IV induction treatment with ustekinumab on a weight-tiered basis at a dose of approximately 6 milligram per kilogram (mg/kg) IV. At Week 8, all participants will receive a 90 mg SC injection of ustekinumab. During the routine care maintenance treatment period, in case of clinical worsening reported by the participant, consistent with disease flare in the investigator's judgment, clinical assessments of disease flare will be performed at the investigator's discretion.

SUMMARY:
The purpose of this study is to evaluate the efficacy of a treat to target strategy coupled with early endoscopic assessment versus a clinically driven (routine care) approach in achieving endoscopic response.

DETAILED DESCRIPTION:
Study investigates benefit of treat to target maintenance treatment strategy versus routine care to test hypothesis that 'treat to target' ustekinumab (UST) maintenance treatment strategy coupled with early endoscopic assessment will result in higher endoscopic response rate after 48 weeks of treatment, compared to pragmatic maintenance treatment strategy. It consists of screening (5 weeks); treatment period (Week 0 to 48); extension period (Weeks 48 to 104) and safety follow up visit (16 weeks after last dose). Participants will be given an option to enter ultrasound sub-study to assess intestinal ultrasound (IUS) parameters indicating transmural changes in response to treatment with UST in participants with Crohn's disease. Study treatment will be unaffected by participation in sub-study which is optional for participants of main study.

ELIGIBILITY:
Inclusion Criteria:

Main Study:

* Have active, moderate to severe, ileal and/or colonic Crohn's disease, demonstrated by: baseline CDAI score of greater than or equal to (>=) 220 and less than equal to (<=) 450, and endoscopy with evidence of active Crohn's disease (defined as simple endoscopic score for Crohn's disease [SES-CD] score >=3 excluding the contribution of the narrowing component score) obtained within the 5 week screening period. A prior endoscopy may be used only if obtained within 3 months prior to baseline (Week 0), in which case the prior endoscopy must be centrally read again and SES-CD calculated based on this second, centralized read-out
* Has had an inadequate response with, lost response to, was intolerant to, or had medical contraindications to either conventional therapy, or one previous biologic therapy approved for the treatment of Crohn's disease in the countries in which the study is conducted
* Are eligible according to tuberculosis (TB) infection screening criteria
* Must sign an informed consent form (ICF) or their legally acceptable representative if applicable must sign) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study.

Sub-study:

* Be enrolled into the main study at a participating site
* Sign a separate ICF indicating that they understand the purpose of and procedures required for this sub-study and are willing to participate in the sub-study
* Satisfy all inclusion criteria and none of the exclusion criteria specified in the main study

Exclusion Criteria:

Main Study:

* Has complications of Crohn's disease such as symptomatic strictures or stenoses, short gut syndrome, or any other manifestation that might be anticipated to require surgery, could preclude the use of the Crohn's Disease Activity Index (CDAI) to assess response to therapy, or would possibly confound the ability to assess the effect of treatment with ustekinumab
* Currently has or is suspected to have an abscess. Recent cutaneous and perianal abscesses are not exclusionary if drained and adequately treated at least 3 weeks prior to baseline, or 8 weeks prior to baseline for intra-abdominal abscesses, provided there is no anticipated need for any further surgery. Participants with active fistulas may be included if there is no anticipation of a need for surgery and there are currently no abscesses identified
* Has had any kind of bowel resection within 6 months prior to baseline
* Has a draining (i.e, functioning) stoma or ostomy
* Has received more than one previous biologic therapy approved for the treatment of Crohn's disease in the countries in which the study is conducted

Sub-study:

* Obesity or other characteristics considered likely to preclude intestinal ultrasound (IUS) visualization of the affected bowel segment
* Normal bowel wall thickness (BWT) (that is, <=2.0 millimeter [mm] for the terminal ileum; <=3.0 mm for the colon) for all bowel segments at baseline (Week 0)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2021-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Cilag Ltd. Clinical Trial, Study Director — Janssen-Cilag Ltd.
Locations (107):
- Belgium (13):
  - GZA Ziekenhuizen, Antwerp
  - Imelda Ziekenhuis, Bonheiden
  - UZ Brussel, Brussels
  - Cliniques Universitaires Saint Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - AZ Maria Middelares, Ghent
  - UZ Gent, Ghent
  - Az Groeninge, Kortrijk
  - UZ Leuven, Leuven
  - CHC MontLegia, Liège
  - CHU de Liege, Liège
  - Algemeen Ziekenhuis Jan Palfijn Merksem, Merksem
  - AZ Damiaan, Ostend
- Czechia (6):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Hepato-gastroenterologie HK, s.r.o., Hradec Králové
  - EGK s.r.o. - Sanatorium sv. Anny, Prague
  - AXON Clinical s.r.o., Prague
  - MEDIENDO s.r.o., Prague
  - ISCARE a.s., Prague
- Denmark (6):
  - Aalborg University Hospital, Aalborg
  - Aarhus Kommunehospital, Aarhus C
  - Abdominalcenter K, København NV
  - Odense Universitetshospital, Odense
  - Silkeborg Hospital, Silkeborg
  - Vejle Sygehus, Vejle
- France (12):
  - Hopital Beaujon, Clichy
  - CHU Grenoble, La Tronche
  - Hopital de Bicetre, Le Kremlin-Bicêtre
  - Hopital Claude Huriez, Lille
  - CHU Saint Eloi, Montpellier
  - CHU de Nice Hopital de l Archet, Nice
  - Hopital Saint Louis, Paris
  - CHU Bordeaux, Pessac
  - Hospices Civils de Lyon HCL, Pierre-Bénite
  - CHU Saint Etienne, Saint-Priest-en-Jarez
  - CHU Rangueil, Toulouse
  - CHU-Nancy, Vandœuvre-lès-Nancy
- Germany (6):
  - Charite Universitatsmedizin Berlin Campus Virchow Klinikum, Berlin
  - Agaplesion Frankfurter Diakonie Kliniken GmbH, Markus Krankenhaus, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
  - Staedtisches Klinikum Lueneburg, Lüneburg
  - Universitaetsklinikum Mannheim, Mannheim
  - MVZ Portal10, Münster
- Italy (13):
  - Policlinico di Bari Ospedale Giovanni XXIII, Bari
  - Policlinico Sant'Orsola Malpighi, Bologna
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - ASST Fatebenefratelli Sacco, Milan
  - Ospedale Classificato Equiparato Sacro Cuore Don Calabria di Negrar, Negrar (VR)
  - Ospedale Villa Sofia-Cervello, Palermo
  - Azienda Ospedaliera G.Salvini Ospedale di Rho, Rho
  - Azienda Ospedaliera San Camillo - Roma, Roma
  - Fondazione Policlinico Gemelli Università Cattolica, Roma
  - Istituto Clinico Humanitas, Rozzano
  - IRCCS Policlinico San Donato, San Donato Milanese
  - AO Ordine Mauriziano, Torino
  - Azienda Sanitaria Universitaria Integrata di Udine, Udine
- Netherlands (6):
  - Meander Medisch Centrum, Amersfoort
  - AMC, Amsterdam
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Rivas Zorggroep, Beatrixziekenhuis, Gorinchem
  - UMCG, Groningen
  - Erasmus MC, Rotterdam
- Portugal (7):
  - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - Centro Hospitalar e Universitário do Algarve, Faro
  - Centro Hospitalar Lisboa Central, EPE - Hospital Santo Antonio dos Capuchos, Lisbon
  - Centro Hospitalar Lisboa Norte EPE Hosp. Santa Maria, Lisbon
  - Centro Hospitalar do Porto, EPE, Porto
  - Centro Hospitalar de Sao Joao Epe, Porto
  - Centro Hospitalar de Tondela Viseu, EPE, Viseu
- Slovakia (7):
  - FNsP F.D.R. Banska Bystrica, Banská Bystrica
  - Gastroenterology Department GASTROMART s.r.o., Bardejov
  - Gastroenterology Center ASSIDUO, Bratislava
  - University Hospital in Bratislava, St. Cyril and Method Hospital, Bratislava
  - KM Management spol. s r.o., Nitra
  - GASTRO I. s.r.o., Prešov
  - Gastroenterology Department ENDOMED, s.r.o., Vranov nad Topľou
- Spain (15):
  - Hosp. Gral. Univ. de Alicante, Alicante
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp Reina Sofia, Córdoba
  - Hosp. Arquitecto Marcide, Ferrol
  - Hosp. Univ. de Bellvitge, L'Hospitalet de Llobregat
  - Hosp. Univ. de La Princesa, Madrid
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp. de Manises, Manises
  - Hosp. Univ. Son Espases, Palma de Mallorca
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. Clinico Univ. de Valencia, Valencia
  - Hosp. Univ. I Politecni La Fe, Valencia
  - Hosp. Clinico Univ. Lozano Blesa, Zaragoza
- Sweden (4):
  - Skane University Hospital, Lund
  - Karolinska University Hospital, Solna
  - Medicinkliniken, Stockholm
  - Danderyd Hospital, Stockholm
- United Kingdom (12):
  - Royal Victoria Hospital, Belfast
  - County Durham and Darlington NHS Foundation Trust, Darlington
  - Ninewells Hospital, Dundee
  - Glasgow Royal Infirmary, Glasgow
  - Royal London Hospital, London
  - Guys St Thomas Hospital, London
  - Kings College Hospital NHS Trust, London
  - St George's University Hospital NHS Foundation Trust, London
  - Whiston Hospital, Prescot
  - Salford Royal NHS Foundation Trust, Salford
  - Southampton University Hospital, Southampton
  - Musgrove Park Hospital, Taunton

REFERENCES:
- [Derived] Hasskamp J, Meinhardt C, Timmer A. Anti-IL-12/23p40 antibodies for induction of remission in Crohn's disease. Cochrane Database Syst Rev. 2025 May 13;5(5):CD007572. doi: 10.1002/14651858.CD007572.pub4. PMID 40357993
- [Derived] Peyrin-Biroulet L, Vermeire S, D'Haens G, Panes J, Dignass A, Magro F, Nazar M, Le Bars M, Lahaye M, Ni L, Bravata I, Lavie F, Daperno M, Lukas M, Armuzzi A, Lowenberg M, Gaya DR, Danese S. Clinical trial: Clinical and endoscopic outcomes with ustekinumab in patients with Crohn's disease: Results from the long-term extension period of STARDUST. Aliment Pharmacol Ther. 2024 Jan;59(2):175-185. doi: 10.1111/apt.17751. Epub 2023 Nov 30. PMID 38036946
- [Derived] Kucharzik T, Wilkens R, D'Agostino MA, Maconi G, Le Bars M, Lahaye M, Bravata I, Nazar M, Ni L, Ercole E, Allocca M, Machkova N, de Voogd FAE, Palmela C, Vaughan R, Maaser C; STARDUST Intestinal Ultrasound study group. Early Ultrasound Response and Progressive Transmural Remission After Treatment With Ustekinumab in Crohn's Disease. Clin Gastroenterol Hepatol. 2023 Jan;21(1):153-163.e12. doi: 10.1016/j.cgh.2022.05.055. Epub 2022 Jul 14. PMID 35842121
- [Derived] Danese S, Vermeire S, D'Haens G, Panes J, Dignass A, Magro F, Nazar M, Le Bars M, Lahaye M, Ni L, Bravata I, Lavie F, Daperno M, Lukas M, Armuzzi A, Lowenberg M, Gaya DR, Peyrin-Biroulet L; STARDUST study group. Treat to target versus standard of care for patients with Crohn's disease treated with ustekinumab (STARDUST): an open-label, multicentre, randomised phase 3b trial. Lancet Gastroenterol Hepatol. 2022 Apr;7(4):294-306. doi: 10.1016/S2468-1253(21)00474-X. Epub 2022 Feb 1. PMID 35120656

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 500 enrolled participants who received at least 1 dose of study medication, 498 participants were included in the analysis because study team decided to exclude one site due to compliance issue. Hence, number of participants who received at least one dose of study medication reduced from 500 to 498 participants.
Groups:
- Induction Period: Ustekinumab (6 Milligrams [mg]/Kilogram [kg]): Participants were administered with approximately 6 mg/kg intravenous (IV) injection of ustekinumab at Week 0 and 90 mg subcutaneous (SC) injection of ustekinumab at Week 8. At Week 16, participants who did not achieve a Crohn's Disease Activity Index (CDAI) improvement (non-responders) of greater than or equal to (>=) 70 points versus Week 0 (CDAI-70), left the study. Participants who achieved CDAI improvement (responders) of at least 70 points versus Week 0 were randomized in open-label maintenance period either in treat to target arm or routine care arm.
- Maintenance Period: Treat to Target: Participants with less than (<) 25 percent (%) improvement in simple endoscopic score for Crohn's disease (SES-CD) at Week 16 versus baseline received ustekinumab 90 mg SC dose 8-weekly maintenance treatment while participants with >= 25% improvement in SES-CD score at Week 16 versus baseline received ustekinumab 90 mg SC dose 12-weekly treatment based on centrally-read ileocolonoscopy findings. From Week 24, participants assigned to the 8-weekly regimen or from Week 20 for the 12-weekly regimen group ustekinumab 90 mg SC maintenance treatment was directed by treat to target assessments based on C-reactive protein (CRP) and CDAI assessments. Participants previously on 12-weekly regimens were adjusted to 8-weekly dosing; those previously on 8-weekly regimens were adjusted to 4-weekly dosing. Participants subsequently failing to meet treatment targets at the next assessment visit 4 weeks after dosing were not able to optimize dosing further and left the study.
- Maintenance Period: Routine Care: Participants received ustekinumab 90 mg SC dose every 8 weeks or every 12 weeks according to clinical judgment. At Week 16, (that is, 8 weeks after the first SC dose), participants who did not show adequate response based on the investigator's judgment received a second ustekinumab 90 mg SC dose at that time. Clinical assessments in case of disease flare were performed at investigator's discretion. Participants who lost response during 12-weekly could adjust the dosing to 8-weekly maintenance treatment. Participants who previously received 8-weekly ustekinumab treatment were unable to adjust the dose following disease flare and left the study as per investigator's judgment.
- Extension Period: Treat to Target: From Week 48, participants continued to receive SC ustekinumab 90 mg in the long-term extension (LTE) period up to Week 104. The frequency of ustekinumab dosing with escalation/de-escalation between once in 12 weeks (q12w)/q8w/q4w was based on the following targets: endoscopic remission (CD [SES-CD] score <=2) and corticosteroid (CS)-free clinical remission (CDAI score of <150 points of >=16 weeks duration) at Week 48; and later, on CS-free clinical remission and biomarker remission (C-reactive protein <=10 milligrams per liter [mg/L] and fecal calprotectin <=250 micrograms per gram [mcg/g]) at 2 consecutive visits 8 weeks apart. Participants on q4w dosing failing to reach targets were discontinued.
- Extension Period: Routine Care: From Week 48, participants continued to receive SC ustekinumab 90 mg in the long-term extension (LTE) period up to Week 104. The frequency of ustekinumab dosing with escalation/de-escalation between once in 12 weeks (q12w)/q8w/q4w was based on the following targets: endoscopic remission (CD [SES-CD] score <=2) and corticosteroid (CS)-free clinical remission (CDAI score of <150 points of >=16 weeks duration) at Week 48; and later, on CS-free clinical remission and biomarker remission (C-reactive protein <=10 mg/L and fecal calprotectin <=250 mcg/g) at 2 consecutive visits 8 weeks apart. Participants on q4w dosing failing to reach targets were discontinued.
Period: Induction Period (16 Weeks)
Arm/Group | Induction Period: Ustekinumab (6 Milligrams [mg]/Kilogram [kg]) | Maintenance Period: Treat to Target | Maintenance Period: Routine Care | Extension Period: Treat to Target | Extension Period: Routine Care
Started | 498 | 0 | 0 | 0 | 0
Participants Who Entered the Maintenance Period | 0 | 219 | 221 | 0 | 0
Participants Who Entered the Extension Period | 0 | 0 | 0 | 147 | 176
Completed | 488 | 0 | 0 | 0 | 0
Not Completed | 10 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 0 | 0
Period: Maintenance Period (Week 16-Week 48)
Arm/Group | Induction Period: Ustekinumab (6 Milligrams [mg]/Kilogram [kg]) | Maintenance Period: Treat to Target | Maintenance Period: Routine Care | Extension Period: Treat to Target | Extension Period: Routine Care
Started | 0 | 219 | 221 | 0 | 0
Completed | 0 | 173 | 193 | 0 | 0
Not Completed | 0 | 46 | 28 | 0 | 0
Not completed — Adverse Event | 0 | 6 | 10 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 2 | 0 | 0
Not completed — Progressive disease | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 21 | 8 | 0 | 0
Not completed — Death | 0 | 2 | 0 | 0 | 0
Not completed — Disease relapse | 0 | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 1 | 0 | 0
Not completed — Received a disallowed concomitant treatment | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 12 | 4 | 0 | 0
Period: Extension Period (Week 48- Week 104)
Arm/Group | Induction Period: Ustekinumab (6 Milligrams [mg]/Kilogram [kg]) | Maintenance Period: Treat to Target | Maintenance Period: Routine Care | Extension Period: Treat to Target | Extension Period: Routine Care
Started | 0 | 0 | 0 | 147 | 176
Completed | 0 | 0 | 0 | 119 | 139
Not Completed | 0 | 0 | 0 | 28 | 37
Not completed — Adverse Event | 0 | 0 | 0 | 10 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 8 | 9
Not completed — Death | 0 | 0 | 0 | 0 | 1
Not completed — Disease relapse | 0 | 0 | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 2
Not completed — Pregnancy | 0 | 0 | 0 | 2 | 4
Not completed — Did not re-consent to protocol amendment 3 | 0 | 0 | 0 | 0 | 1
Not completed — Non-compliance with study drug | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 5 | 9

BASELINE CHARACTERISTICS:
Arm/Group | Induction Period: Ustekinumab (6 Milligrams [mg]/Kilogram [kg])
Number analyzed (Participants) | 498
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (12.96) [lower limit 12.96]
Age, Customized [Count of Participants; unit: Participants]
  18-25 years | 112
  26-50 years | 302
  51-64 years | 71
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 257
  Male | 241
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 29
  Czech Republic | 24
  Denmark | 15
  France | 51
  Germany | 26
  Italy | 166
  Netherlands | 19
  Portugal | 37
  Slovakia | 30
  Spain | 47
  Sweden | 15
  United Kingdom | 39

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Endoscopic Response at Week 48
Description: Endoscopic response defined as showing a reduction from baseline in simple endoscopic score for Crohn's disease (SES-CD) of greater than or equal to (>=) 50 percent (%). SES-CD is a validated instrument reflecting an endoscopist global appraisal of mucosal lesions in Crohn's disease. SES-CD grades lesions by location (5 bowel segments: ileum, right colon, transverse colon, left colon, and rectum) using 4 endoscopic variables: ulcer size, extent of ulcerated surface, extent of affected surface, and presence/type of narrowing. Total SES-CD is sum of 4 variables for all 5 bowel segments. Scores range from 0-60 with higher scores indicating more severe disease. Randomized participants who stopped treatment before reaching Week 48 due to any reason, or participants without endoscopic data at Week 48 were analyzed as nonresponders.
Time Frame: Week 48
Population: Full randomized analysis set (FRAS) included all participants who received at least 1 dose of study agent and were randomized at Week 16, regardless of study treatment being administered once randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Maintenance Period: Treat to Target | Maintenance Period: Routine Care
Number analyzed (Participants) | 219 | 221
Percentage of Participants | 37.9 (31.4) [31.4 to 44.7] | 29.9 (23.9) [23.9 to 36.4]
Statistical Analysis 1: Comparison: Maintenance Period: Treat to Target vs Maintenance Period: Routine Care; Test type: Superiority; p = 0.0871, Cochran-Mantel-Haenszel

2. Secondary Outcome: Percentage of Participants With Endoscopic Response at Week 48 (Premature Drop-outs Excluded)
Description: Endoscopic response defined as showing a reduction from baseline in SES-CD (a validated instrument reflecting an endoscopist's global appraisal of mucosal lesions) score of >=50%. SES-CD grades lesions by location (5 bowel segments: ileum, right colon, transverse colon, left colon, and rectum) using 4 endoscopic variables: ulcer size, extent of ulcerated surface, extent of affected surface, and presence/type of narrowing. Total SES-CD is calculated as sum of 4 variables for 5 bowel segments. Scores ranges 0-60. Higher scores indicates more severe disease. Randomized participants who stopped treatment before reaching Week 48 due to reasons other than lack/loss of efficacy were excluded from analysis.
Time Frame: Week 48
Population: FRAS included all participants who received at least 1 dose of study agent and were randomized at Week 16, regardless of study treatment being administered once randomized. Here, 'N' (Number of participants analyzed) included participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Maintenance Period: Treat to Target | Maintenance Period: Routine Care
Number analyzed (Participants) | 193 | 198
Percentage of Participants | 43.0 (35.9) [35.9 to 50.3] | 32.3 (25.9) [25.9 to 39.3]

3. Secondary Outcome: Percentage of Participants With Endoscopic Response at Week 48 (Last Observation Carried Forward [LOCF])
Description: Endoscopic response defined as a reduction from baseline in SES-CD score of >= 50%. SES-CD is a validated instrument reflecting an endoscopist global appraisal of mucosal lesions in Crohn's disease. SES-CD grades lesions by location (5 bowel segments: ileum, right colon, transverse colon, left colon, and rectum) using 4 endoscopic variables: ulcer size, extent of ulcerated surface, extent of affected surface, and presence/type of narrowing. The total SES-CD was calculated as the sum of the 4 variables for the 5 bowel segments. Scores range from 0 to 60, with higher scores indicating more severe disease. LOCF: Participants who had a missing value at Week 48 or who stopped treatment before reaching Week 48 had their last non-missing value carried forward.
Time Frame: Week 48 (LOCF)
Population: FRAS included all participants who received at least 1 dose of study agent and were randomized at Week 16, regardless of study treatment being administered once randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Maintenance Period: Treat to Target | Maintenance Period: Routine Care
Number analyzed (Participants) | 219 | 221
Percentage of Participants | 40.2 (33.6) [33.6 to 47.0] | 30.8 (24.8) [24.8 to 37.3]

4. Secondary Outcome: Percentage of Participants With Clinical Response at Weeks 16, 48, and Endpoint (Week 48 [LOCF])
Description: Clinical response defined as a >=100-point reduction from the baseline in Crohn's Disease Activity Index (CDAI) score, or a CDAI score of <150. The CDAI score is used to quantify the symptoms of participants with Crohn's Disease. A decrease in CDAI over time indicates improvement in disease activity. In general, CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities. Participants with missing data were considered as non-responder. LOCF: Participants who had a missing value at Week 48 or who stopped treatment before reaching Week 48 had their last non-missing value carried forward. Endpoint is defined as the last available postbaseline result within the main analysis period (that is, first 48 weeks of the study).
Time Frame: Weeks 16, 48, and Endpoint (Week 48 [LOCF])
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Maintenance Period: Treat to Target | Maintenance Period: Routine Care
Number analyzed (Participants) | 219 | 221
Percentage of Participants
  Week 16 | 84.5 [80.0 to 89.8] | 89.6 [84.8 to 93.3]
  Week 48 | 68.0 [61.4 to 74.2] | 77.8 [71.8 to 83.1]
  Endpoint (Week 48 [LOCF]) | 89.5 [84.7 to 93.2] | 89.6 [84.8 to 93.3]

5. Secondary Outcome: Percentage of Participants With Clinical Remission at Weeks 16, 48, and Endpoint (Week 48 [LOCF])
Description: Clinical Remission defined as a CDAI score of <150 points. The CDAI score is used to quantify the symptoms of participants with Crohn's Disease. A decrease in CDAI over time indicates improvement in disease activity. In general, CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities. Participants with missing data were considered as non-remitter. LOCF: Participants who had a missing value at Week 48 or who stopped treatment before reaching Week 48 had their last non-missing value carried forward. Endpoint is defined as the last available postbaseline result within the main analysis period (that is, first 48 weeks of the study).
Time Frame: Weeks 16, 48, and Endpoint (Week 48 [LOCF])
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Maintenance Period: Treat to Target | Maintenance Period: Routine Care
Number analyzed (Participants) | 219 | 221
Percentage of Participants
  Week 16 | 72.1 [65.7 to 78.0] | 74.2 [67.9 to 79.8]
  Week 48 | 61.6 [54.9 to 68.1] | 69.7 [63.2 to 75.7]
  Endpoint (Week 48 [LOCF]) | 77.2 [71.0 to 82.6] | 78.3 [72.3 to 83.5]

6. Secondary Outcome: Percentage of Participants With Endoscopic Remission at Weeks 16, 48, and Endpoint (Week 48 [LOCF])
Description: Percentage of participants with Endoscopic remission defined as SES-CD score <=2 at Weeks 16, 48, and Endpoint (Week 48 [LOCF]) were reported. SES-CD is a validated instrument reflecting an endoscopist global appraisal of mucosal lesions in Crohn's disease. SES-CD grades lesions by location (5 bowel segments: ileum, right colon, transverse colon, left colon, and rectum) using 4 endoscopic variables: ulcer size, extent of ulcerated surface, extent of affected surface, and presence/type of narrowing. Total SES-CD is sum of 4 variables for all 5 bowel segments. Scores range from 0-60 with higher scores indicating more severe disease. LOCF: Participants who had a missing value at Week 48 or who stopped treatment before reaching Week 48 had their last non-missing value carried forward. Endpoint is defined as the last available postbaseline result within the main analysis period (that is, first 48 weeks of the study).
Time Frame: Weeks 16, 48, and Endpoint (Week 48 [LOCF])
Population: FRAS included all participants who received at least 1 dose of study agent and were randomized at Week 16, regardless of study treatment being administered once randomized. Here, 'n' (number analyzed) refers participants analyzed at specified timepoints. Data was not collected for routine care arm at Week 16 as per planned analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Maintenance Period: Treat to Target | Maintenance Period: Routine Care
Number analyzed (Participants) | 219 | 221
Percentage of Participants
  Week 16: number analyzed (Participants) | 219 | 0
  Week 16 | 11.4 [7.5 to 16.4] |
  Week 48 | 11.4 [7.5 to 16.4] | 14.5 [10.1 to 19.8]
  Endpoint (Week 48 [LOCF]) | 11.9 [7.9 to 16.9] | 15.4 [10.9 to 20.8]

7. Secondary Outcome: Percentage of Participants With Mucosal Healing at Weeks 16, 48, and Endpoint (Week 48 [LOCF])
Description: Mucosal healing is defined as the complete absence of mucosal ulcerations in any ileocolonic segment. SES-CD grades lesions by location (5 bowel segments: ileum, right colon, transverse colon, left colon, and rectum) using 4 endoscopic variables: ulcer size, extent of ulcerated surface, extent of affected surface, and presence/type of narrowing. Total SES-CD is sum of 4 variables for all 5 bowel segments. Scores range from 0-60 with higher scores indicating more severe disease. LOCF: Participants who had a missing value at Week 48 or who stopped treatment before reaching Week 48 had their last non-missing value carried forward. Endpoint is defined as the last available postbaseline result within the main analysis period (i.e. first 48 weeks of the study).
Time Frame: Weeks 16, 48, and Endpoint (Week 48 [LOCF])
Population: FRAS included all participants who received at least 1 dose of study agent and were randomized at Week 16, regardless of study treatment being administered once randomized. Here, 'n' (number analyzed) is defined as number of participants who were analyzed at specified timepoints. Data was not collected for routine care arm at Week 16 as per planned analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Maintenance Period: Treat to Target | Maintenance Period: Routine Care
Number analyzed (Participants) | 219 | 221
Percentage of Participants
  Week 16: number analyzed (Participants) | 219 | 0
  Week 16 | 16.0 [11.4 to 21.5] |
  Week 48 | 14.2 [9.8 to 19.5] | 16.7 [12.1 to 22.3]
  Endpoint (Week 48 [LOCF]) | 14.6 [10.2 to 20.0] | 17.6 [12.9 to 23.3]

8. Secondary Outcome: Percentage of Participants With Corticosteroid-free Clinical Remission at Week 48 and Endpoint (Week 48 [LOCF])
Description: Corticosteroid-free Clinical Remission at Week 48 and Endpoint (Week 48 [LOCF]) is defined as a CDAI score <150 and not taking any corticosteroids for at least 30 days prior to Week 48 and Endpoint assessment. The CDAI score is used to quantify the symptoms of participants with Crohn's Disease. A decrease in CDAI over time indicates improvement in disease activity. In general, CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities. Participants with missing data were analyzed as non-remitter. LOCF: Participants who had a missing value at Week 48 or who stopped treatment before reaching Week 48 had their last non-missing value carried forward. Endpoint is defined as the last available postbaseline result within the main analysis period (that is, first 48 weeks of the study).
Time Frame: Week 48 and Endpoint (Week 48 [LOCF])
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Maintenance Period: Treat to Target | Maintenance Period: Routine Care
Number analyzed (Participants) | 219 | 221
Percentage of Participants
  Week 48 | 56.6 [49.8 to 63.3] | 63.3 [56.6 to 69.7]
  Endpoint (Week 48 [LOCF]) | 70.8 [64.3 to 76.7] | 69.7 [63.2 to 75.7]

9. Secondary Outcome: Percentage of Participants With Corticosteroid-free Endoscopic Response at Weeks 16, 48, and Endpoint (Week 48 [LOCF])
Description: Corticosteroid-free endoscopic response defined as a reduction from baseline in SES-CD score of >=50% and not taking any corticosteroids for at least 30 days prior to Weeks 16, 48 and endpoint (Week 48 [LOCF]). SES-CD grades lesions by location (5 bowel segments: ileum, right colon, transverse colon, left colon, and rectum) using 4 endoscopic variables: ulcer size, extent of ulcerated surface, extent of affected surface, and presence/type of narrowing. Total score is sum of 4 variables. Scores range 0-60. Higher scores means severe disease. Participants with missing data were analyzed as No SES-CD Improvement. LOCF: Participants who had a missing value at Week 48 or who stopped treatment before reaching Week 48 had their last non-missing value carried forward. Endpoint defined as last available postbaseline result within main analysis period (i.e., first 48 weeks).
Time Frame: Weeks 16, 48, and Endpoint (Week 48 [LOCF])
Population: FRAS included all participants who received at least 1 dose of study agent and were randomized at Week 16, regardless of study treatment being administered once randomized. Here, 'n' (number analyzed) included participants analyzed at specified timepoints. Data was not collected for routine care arm at Week 16 as per planned analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Maintenance Period: Treat to Target | Maintenance Period: Routine Care
Number analyzed (Participants) | 219 | 221
Percentage of Participants
  Week 16: number analyzed (Participants) | 219 | 0
  Week 16 | 26.5 [20.8 to 32.9] |
  Week 48 | 33.8 [27.6 to 40.5] | 28.5 [22.7 to 34.9]
  Endpoint (Week 48 [LOCF]) | 36.1 [29.7 to 42.8] | 29.4 [23.5 to 35.9]

10. Secondary Outcome: Change From Baseline in Serum C-reactive Protein (CRP)
Description: Change from baseline in serum CRP were reported. LOCF: Participants who had a missing value at Week 48 or who stopped treatment before reaching Week 48 had their last non-missing value carried forward. Endpoint is defined as the last available postbaseline result within the main analysis period (that is, first 48 weeks of the study).
Time Frame: Baseline, Weeks 16, 48 and Endpoint (Week 48 [LOCF]
Population: FRAS included all participants who received at least 1 dose of study agent and were randomized at Week 16, regardless of study treatment being administered once randomized. Here, 'N' (Number analyzed) included participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Milligrams per liter (mg/L)
Arm/Group | Maintenance Period: Treat to Target | Maintenance Period: Routine Care
Number analyzed (Participants) | 218 | 219
Milligrams per liter (mg/L)
  Change at Week 16 | -7.717 (22.0246) | -7.345 (17.5658)
  Change at Week 48 | -7.839 (22.6777) | -7.909 (22.2139)
  Change at Endpoint (Week 48 [LOCF]) | -7.839 (22.6777) | -7.909 (22.2139)

11. Secondary Outcome: Change From Baseline in Fecal Calprotectin (FC)
Description: Change from baseline in FC were reported. LOCF: Participants who had a missing value at Week 48 or who stopped treatment before reaching Week 48 had their last non-missing value carried forward. Endpoint is defined as the last available postbaseline result within the main analysis period (that is, first 48 weeks of the study).
Time Frame: Baseline, Weeks 16, 48 and Endpoint (Week 48 [LOCF])
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micrograms per gram (mcg/g)
Arm/Group | Maintenance Period: Treat to Target | Maintenance Period: Routine Care
Number analyzed (Participants) | 196 | 189
Micrograms per gram (mcg/g)
  Change at Week 16 | -988.8 (3243.61) | -728.2 (2238.60)
  Change at Week 48 | -1191.6 (3441.64) | -744.4 (2589.30)
  Change at Endpoint (Week 48 [LOCF]) | -1191.6 (3441.64) | -744.4 (2589.30)

12. Secondary Outcome: Percentage of Participants With Inflammatory Bowel Disease Questionnaire (IBDQ) Response
Description: IBDQ response was defined as >= 16-point improvement in IBDQ total score from baseline. The IBDQ is 32-item questionnaire for participants with IBD used to evaluate disease-specific health-related quality of life. Each item score ranged from 1 (worst possible response) to 7 (best possible response). Each items were grouped into 4 domains: bowel function, emotional status, systemic symptoms and social function. The 4 domains were scored as: 10 to 70 (bowel symptoms); 5 to 35 (systemic symptoms); 12 to 84 (emotional function); 5 to 35 (social function). For each domain, higher score indicated better quality of life. Total score is sum of each item score and ranges from 32 to 224 with higher score indicating better quality of life. LOCF: Participants who had a missing value at Week 48 or who stopped treatment before reaching Week 48 had their last non-missing value carried forward. Endpoint defined as last available postbaseline result within main analysis period (i.e, first 48 weeks).
Time Frame: Weeks 16, 48, and Endpoint (Week 48 [LOCF])
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Maintenance Period: Treat to Target | Maintenance Period: Routine Care
Number analyzed (Participants) | 219 | 221
Percentage of Participants
  Week 16 | 71.7 [65.2 to 77.6] | 75.1 [68.9 to 80.7]
  Week 48 | 58.4 [51.6 to 65.0] | 67.0 [60.3 to 73.1]
  Endpoint (Week 48 [LOCF]) | 77.2 [71.0 to 82.6] | 77.8 [71.8 to 83.1]

13. Secondary Outcome: Percentage of Participants With 7-point Change From Baseline in Work Productivity and Activity Impairment (WPAI) Scores for Each Domain
Description: Percentage of participants with 7-point change from baseline in WPAI scores for each domain were reported. WPAI is 6-item (7-day recall period) well-validated questionnaire to measure impairments in work and activities that produces 4 types of domains: absenteeism (work time missed), presenteeism (impairment at work/reduced on-the-job effectiveness), work productivity loss (overall work impairment/absenteeism plus presenteeism), activity impairment. Participants who answered first question of the questionnaire 'Are you currently employed' as 'Yes' were included in absenteeism, presenteeism, and work productivity. In activity impairment all participants were included. Each score range: 0-100, higher scores=greater impairment and less productivity. LOCF: Participants who had missing value at Week 48 or stopped treatment before reaching Week 48 had last non-missing value carried forward. Endpoint: last available postbaseline result in main analysis period (first 48 weeks).
Time Frame: Weeks 16, 48, and Endpoint (Week 48 [LOCF])
Population: FRAS included all participants who received at least 1 dose of study agent and were randomized at Week 16, regardless of study treatment being administered once randomized. Here, 'N' (Number of participants analyzed) included participants who were evaluable for this outcome measure. Here, 'n' (number analyzed) is defined as participants analyzed for specified categories.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Maintenance Period: Treat to Target | Maintenance Period: Routine Care
Number analyzed (Participants) | 212 | 215
Percentage of Participants
  Week 16: Absenteeism: number analyzed (Participants) | 86 | 96
  Week 16: Absenteeism | 34.9 [24.9 to 45.9] | 39.6 [29.7 to 50.1]
  Week 48: Absenteeism: number analyzed (Participants) | 60 | 77
  Week 48: Absenteeism | 35.0 [23.1 to 48.4] | 36.4 [25.7 to 48.1]
  Endpoint (Week 48 [LOCF]): Absenteeism: number analyzed (Participants) | 83 | 81
  Endpoint (Week 48 [LOCF]): Absenteeism | 34.9 [24.8 to 46.2] | 36.3 [26.4 to 47.0]
  Week 16: Presenteeism: number analyzed (Participants) | 105 | 104
  Week 16: Presenteeism | 70.5 [60.8 to 79.0] | 76.9 [67.6 to 84.6]
  Week 48: Presenteeism: number analyzed (Participants) | 78 | 92
  Week 48: Presenteeism | 73.1 [61.8 to 82.5] | 72.8 [62.6 to 81.6]
  Endpoint (Week 48 [LOCF]): Presenteeism: number analyzed (Participants) | 102 | 106
  Endpoint (Week 48 [LOCF]): Presenteeism | 69.6 [59.7 to 78.3] | 69.8 [60.1 to 78.3]
  Week 16: Work Productivity Loss: number analyzed (Participants) | 77 | 82
  Week 16: Work Productivity Loss | 71.4 [60.0 to 81.2] | 70.7 [59.6 to 80.3]
  Week 48: Work Productivity Loss: number analyzed (Participants) | 56 | 48
  Week 48: Work Productivity Loss | 75.0 [61.6 to 85.6] | 72.1 [59.9 to 82.3]
  Endpoint (Week 48 [LOCF]): Work Productivity Loss: number analyzed (Participants) | 76 | 79
  Endpoint (Week 48 [LOCF]): Work Productivity Loss | 72.4 [60.9 to 82.0] | 69.6 [58.2 to 79.5]
  Week 16: Activity Impairment: number analyzed (Participants) | 204 | 207
  Week 16: Activity Impairment | 72.1 [65.4 to 78.1] | 78.3 [72.0 to 83.7]
  Week 48: Activity Impairment: number analyzed (Participants) | 156 | 178
  Week 48: Activity Impairment | 74.4 [66.8 to 81.0] | 71.9 [64.7 to 78.4]
  Endpoint (Week 48 [LOCF]): Activity Impairment | 67.9 [61.2 to 74.2] | 70.7 [64.1 to 76.7]

14. Secondary Outcome: Change From Baseline in IBDQ Score
Description: The IBDQ is 32-item questionnaire used to evaluate disease-specific health-related quality of life. Each item score ranged from 1 (worst possible response) to 7 (best possible response). Items were grouped into 4 domains: bowel function, emotional status, systemic symptoms and social function with scored as follows: 10 to 70 (bowel symptoms); 5 to 35 (systemic symptoms); 12 to 84 (emotional function); and 5 to 35 (social function). Higher score, better quality of life. Total score is sum of each item score and ranges from 32 to 224. LOCF: Participants who had a missing value at Week 48 or who stopped treatment before reaching Week 48 had their last non-missing value carried forward. Endpoint defined as last available postbaseline result within main analysis period (that is, first 48 weeks of the study). Only participants with non-missing baseline value and at least one non-missing post-baseline value during main treatment period were included in analysis.
Time Frame: Baseline, Weeks 16, 48, and Endpoint (Week 48 [LOCF])
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Maintenance Period: Treat to Target | Maintenance Period: Routine Care
Number analyzed (Participants) | 214 | 217
Units on a scale
  Change at Week 16 | 41.3 (34.24) | 44.7 (33.20)
  Change at Week 48 | 43.7 (35.16) | 44.3 (36.94)
  Change at Endpoint (Week 48 [LOCF]) | 43.7 (35.16) | 44.3 (36.94)

15. Secondary Outcome: Change From Baseline in European Quality Of Life 5 Dimensions 5 Level (EQ-5D-5L) Visual Analog Scale (VAS) Score
Description: EQ-5D-5L, validated quality-of-life instrument completed by participants. It consists of EQ-5D-5L descriptive system and EQ-VAS. EQ-5D-5L descriptive system comprises 5 dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) describes participants current health state. Each dimension scores where 1 indicates no problems and 5 indicates extreme problems. EQ-5D-5L VAS records the respondent's self-rated, visual analogue scale score on a scale of 0-100, where 0 labelled as 'the worst health you can imagine and 100 labelled 'the best health you can imagine.' LOCF: Participants who had a missing value at Week 48 or who stopped treatment before reaching Week 48 had their last non-missing value carried forward. Endpoint defined as last available postbaseline result within main analysis period (i.e., first 48 weeks).
Time Frame: Baseline, Weeks 16, 48, and Endpoint (Week 48 [LOCF])
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Maintenance Period: Treat to Target | Maintenance Period: Routine Care
Number analyzed (Participants) | 218 | 218
Units on a scale
  Change at Week 16 | 16.7 (20.19) | 18.7 (20.16)
  Change at Week 48 | 16.5 (22.77) | 16.1 (21.71)
  Change at Endpoint (Week 48 [LOCF]) | 16.5 (22.77) | 16.1 (21.71)

16. Secondary Outcome: Changes From Baseline in Functional Assessment of Chronic Illness Therapy-fatigue (FACIT-F) Scale Score
Description: The FACIT-F scale is a 13-item fatigue scale with a 7-day recall period. It measures the level of fatigue during the usual daily activities. The level of fatigue is measured on a 4-point Likert scale (0=very much fatigue to 4=not at all fatigue). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worst score) to 52 (best score). LOCF: Participants who had a missing value at Week 48 or who stopped treatment before reaching Week 48 had their last non-missing value carried forward. Endpoint is defined as the last available postbaseline result within the main analysis period (that is, first 48 weeks of the study).
Time Frame: Baseline, Weeks 16, 48, and Endpoint (Week 48 [LOCF])
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Maintenance Period: Treat to Target | Maintenance Period: Routine Care
Number analyzed (Participants) | 219 | 220
Units on a scale
  Change at Week 16 | 9.1 (10.57) | 11.6 (10.12)
  Change at Week 48 | 9.9 (11.35) | 10.0 (11.11)
  Change at Endpoint (Week 48 [LOCF]) | 9.9 (11.35) | 10.0 (11.11)

17. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) Score
Description: The HADS Score is a validated 14-item scale with 7 of the items relating to anxiety and 7 relating to depression. Each item is scored from 0 to 3, with higher scores indicating greater likelihood of depression or anxiety. Cases of anxiety or depression are each defined by subscale scores of 8 or greater and categorized as normal (score of 0 to 7), mild (score of 8 to 10), moderate (score of 11 to 14), and severe (score of 15 to 21). LOCF: Participants who had a missing value at Week 48 or who stopped treatment before reaching Week 48 had their last non-missing value carried forward. Endpoint is defined as the last available postbaseline result within the main analysis period (that is, first 48 weeks of the study).
Time Frame: Baseline, Weeks 16, 48, and Endpoint (Week 48 [LOCF])
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Maintenance Period: Treat to Target | Maintenance Period: Routine Care
Number analyzed (Participants) | 216 | 217
Units on a scale
  Change at Week 16: Anxiety | -2.5 (3.43) | -2.5 (3.88)
  Change at Week 16: Depression | -2.5 (3.59) | -2.4 (3.41)
  Change at Week 48: Anxiety | -2.5 (3.64) | -2.7 (4.05)
  Change at Week 48: Depression | -2.4 (4.00) | -2.2 (3.97)
  Change at Endpoint (Week 48 [LOCF]): Anxiety | -2.5 (3.64) | -2.7 (4.05)
  Change at Endpoint (Week 48 [LOCF]): Depression | -2.4 (4.00) | -2.2 (3.97)

18. Secondary Outcome: Change From Baseline in WPAI Score
Description: The WPAI questionnaire is a well-validated instrument to measure impairments in work and activities. It is a 6-item questionnaire with a 7-day recall period. The WPAI questionnaire produces 4 types of scores: absenteeism (work time missed), presenteesism (impairment at work/reduced on-the-job effectiveness), work productivity loss (overall work impairment/absenteeism plus presenteeism), and activity impairment. Each score ranges from 0 to 100 with higher scores indicating greater impairment and less productivity. LOCF: Participants who had a missing value at Week 48 or who stopped treatment before reaching Week 48 had their last non-missing value carried forward. Endpoint is defined as the last available postbaseline result within the main analysis period (that is, first 48 weeks of the study).
Time Frame: Baseline, Weeks 16, 48, and Endpoint (Week 48 [LOCF])
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Maintenance Period: Treat to Target | Maintenance Period: Routine Care
Number analyzed (Participants) | 212 | 215
Units on a scale
  Absenteeism: Change at Week 16: number analyzed (Participants) | 86 | 96
  Absenteeism: Change at Week 16 | -12.9 (31.39) | -12.5 (30.86)
  Absenteeism: Change at Week 48: number analyzed (Participants) | 60 | 77
  Absenteeism: Change at Week 48 | -13.9 (34.13) | -14.8 (30.22)
  Absenteeism: Change at Endpoint (Week 48 [LOCF]): number analyzed (Participants) | 83 | 91
  Absenteeism: Change at Endpoint (Week 48 [LOCF]) | -13.0 (34.87) | -12.1 (31.92)
  Presenteeism: Change at Week 16 | -23.3 (27.76) | -26.2 (30.09)
  Presenteeism: Change at Week 48: number analyzed (Participants) | 78 | 92
  Presenteeism: Change at Week 48 | -30.0 (31.83) | -26.0 (28.90)
  Presenteeism: Change at Endpoint (Week 48 [LOCF]): number analyzed (Participants) | 102 | 106
  Presenteeism: Change at Endpoint (Week 48 [LOCF]) | -26.5 (30.50) | -22.5 (30.99)
  Work Productivity Loss: Change at Week 16: number analyzed (Participants) | 77 | 82
  Work Productivity Loss: Change at Week 16 | -25.2 (27.71) | -27.2 (31.79)
  Work Productivity Loss: Change at Week 48: number analyzed (Participants) | 56 | 68
  Work Productivity Loss: Change at Week 48 | -33.0 (33.98) | -28.0 (31.66)
  Work Productivity Loss: Change at Endpoint (Week 48 [LOCF]): number analyzed (Participants) | 76 | 79
  Work Productivity Loss: Change at Endpoint (Week 48 [LOCF]) | -29.1 (32.91) | -24.1 (33.97)
  Activity Impairment: Change at Week 16: number analyzed (Participants) | 156 | 178
  Activity Impairment: Change at Week 16 | -24.1 (27.23) | -27.3 (26.77)
  Activity Impairment: Change at Week 48: number analyzed (Participants) | 156 | 178
  Activity Impairment: Change at Week 48 | -29.2 (29.65) | -24.8 (28.96)
  Activity Impairment: Change at Endpoint (Week 48 [LOCF]) | -25.5 (29.13) | -23.6 (29.08)

19. Secondary Outcome: Change From Baseline in Time Lost From Work
Description: Time lost from work was collected by asking the participants a single question, "How many days did you miss from work due to your Crohn's disease in the last 4 weeks?" LOCF: Participants who had a missing value at Week 48 or who stopped treatment before reaching Week 48 had their last non-missing value carried forward. Endpoint is defined as the last available postbaseline result within the main analysis period (that is, first 48 weeks of the study).
Time Frame: Baseline, Weeks 16, 48, and Endpoint (Week 48 [LOCF])
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Maintenance Period: Treat to Target | Maintenance Period: Routine Care
Number analyzed (Participants) | 133 | 139
Days
  Change at Week 16 | -1.7 (4.32) | -1.8 (6.03)
  Change at Week 48 | -1.8 (4.58) | -2.2 (5.99)
  Change at Endpoint (Week 48 [LOCF]) | -1.8 (4.58) | -2.2 (5.99)

20. Secondary Outcome: Number of Participants With Adverse Events (AEs) That Occurred in Participants Administered With Ustekinumab up to Week 48
Description: An adverse event is any untoward medical event that occurs in participants administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Time Frame: Up to Week 48
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Period: Treat to Target | Maintenance Period: Routine Care
Number analyzed (Participants) | 219 | 221
Participants | 188 | 179

21. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight were reported. LOCF: Participants who had a missing value at Week 48 or who stopped treatment before reaching Week 48 had their last non-missing value carried forward. Endpoint is defined as the last available postbaseline result within the main analysis period (that is, first 48 weeks of the study).
Time Frame: Baseline, Weeks 16, 48, and Endpoint (Week 48 [LOCF])
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Kilograms (Kg)
Arm/Group | Maintenance Period: Treat to Target | Maintenance Period: Routine Care
Number analyzed (Participants) | 219 | 221
Kilograms (Kg)
  Change at Week 16 | 1.56 (2.996) | 1.16 (3.586)
  Change at Week 48 | 2.38 (4.682) | 1.39 (4.877)
  Change at Endpoint (Week 48 [LOCF]) | 2.38 (4.682) | 1.39 (4.877)

22. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Description: Change from baseline in BMI were reported. BMI is a person's weight (in kilograms) divided by the square of height (in meters).LOCF: Participants who had a missing value at Week 48 or who stopped treatment before reaching Week 48 had their last non-missing value carried forward. Endpoint is defined as the last available postbaseline result within the main analysis period (that is, first 48 weeks of the study).
Time Frame: Baseline, Weeks 16, 48, and Endpoint (Week 48 [LOCF])
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Kilograms per meter square (Kg/m^2)
Arm/Group | Maintenance Period: Treat to Target | Maintenance Period: Routine Care
Number analyzed (Participants) | 219 | 221
Kilograms per meter square (Kg/m^2)
  Change at Week 16 | 0.54 (1.052) | 0.37 (1.236)
  Change at Week 48 | 0.82 (1.622) | 0.46 (1.665)
  Change at Endpoint (Week 48 [LOCF]) | 0.82 (1.622) | 0.46 (1.665)

23. Secondary Outcome: Change From Baseline in Blood Pressure
Description: Change from baseline in Blood Pressure (Systolic Blood Pressure [SPB] and Diastolic Blood Pressure [DBP]) were reported. LOCF: Participants who had a missing value at Week 48 or who stopped treatment before reaching Week 48 had their last non-missing value carried forward. Endpoint is defined as the last available postbaseline result within the main analysis period (i.e. first 48 weeks of the study).
Time Frame: Baseline, Weeks 16, 48, and Endpoint (Week 48 [LOCF])
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Maintenance Period: Treat to Target | Maintenance Period: Routine Care
Number analyzed (Participants) | 219 | 221
Millimeter of mercury (mmHg)
  SBP: Change at Week 16 | 2.3 (13.16) | 0.3 (12.59)
  SBP: Change at Week 48 | 1.9 (13.21) | 0.5 (12.47)
  SBP: Change at Endpoint (Week 48 [LOCF]) | 1.9 (13.21) | 0.5 (12.47)
  DBP: Change at Week 16 | 1.1 (9.46) | 0.8 (9.81)
  DBP: Change at Week 48 | 1.2 (10.02) | 0.6 (9.85)
  DBP: Change at Endpoint (Week 48 [LOCF]) | 1.2 (10.02) | 0.6 (9.85)

24. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Change from baseline in pulse rate were reported. LOCF: Participants who had a missing value at Week 48 or who stopped treatment before reaching Week 48 had their last non-missing value carried forward. Endpoint is defined as the last available postbaseline result within the main analysis period (i.e. first 48 weeks of the study).
Time Frame: Baseline, Weeks 16, 48, and Endpoint (Week 48 [LOCF])
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Maintenance Period: Treat to Target | Maintenance Period: Routine Care
Number analyzed (Participants) | 219 | 221
Beats/minute
  Change at Week 16 | -1.5 (11.98) | -2.0 (11.51)
  Change at Week 48 | -0.2 (13.39) | -1.7 (12.16)
  Change at Endpoint (Week 48 [LOCF]) | -0.2 (13.39) | -1.7 (12.16)

ADVERSE EVENTS:
Time Frame: Induction Period= Baseline up to Week 16; Maintenance Period= Baseline up to Week 48; Extension Period/End of Study= Baseline up to Week 104. In maintenance period and extension period AEs are reported that occurred between baseline and Week 48 and between baseline and Week 104, respectively, i.e., there is an overlap.
Description: For Induction period: The safety analysis set included all participants from the full analysis set (FAS). For Maintenance period: Full randomized analysis set (FRAS) included all participants who received at least 1 dose of study agent and were randomized at Week 16, regardless of study treatment being administered once randomized. For Extension period: Modified FAS (mFAS) included all participants randomized at Week 16 that completed Week 48 and entered the extension period.
Groups:
- Induction Period: Participants were administered with approximately 6 mg/kg intravenous (IV) injection of ustekinumab at Week 0 and 90 mg subcutaneous (SC) injection of ustekinumab at Week 8. At Week 16, participants who did not achieve a Crohn's Disease Activity Index (CDAI) improvement (non-responders) of greater than or equal to (>=) 70 points versus Week 0 (CDAI-70), left the study. Participants who achieved CDAI improvement (responders) of at least 70 points versus Week 0 were randomized in open-label maintenance period either with treat to target arm or routine care arm.
Arm/Group | Induction Period | Maintenance Period: Treat to Target | Maintenance Period: Routine Care | Extension Period: Treat to Target | Extension Period: Routine Care
All-Cause Mortality (participants affected / at risk) | 0/498 | 2/219 | 0/221 | 0/147 | 1/176
Serious Adverse Events (participants affected / at risk) | 28/498 | 26/219 | 29/221 | 21/147 | 23/176
Other Adverse Events (participants affected / at risk) | 238/498 | 158/219 | 150/221 | 125/147 | 135/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Period (N=498) | Maintenance Period: Treat to Target (N=219) | Maintenance Period: Routine Care (N=221) | Extension Period: Treat to Target (N=147) | Extension Period: Routine Care (N=176)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina Pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiac Failure Acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 2 (3)
Anal Fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Crohn's Disease (Gastrointestinal disorders) | 6 (7) | 4 (4) | 8 (10) | 1 (1) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fistula of Small Intestine (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal Stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intra-Abdominal Fluid Collection (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large Intestine Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large Intestine Polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Wall Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abscess Intestinal (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anal Abscess (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bartholinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Campylobacter Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Covid-19 Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enteritis Infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Infectious Colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large Intestine Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Perirectal Abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Joint Dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Body Temperature Increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervix Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuroendocrine Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Superficial Spreading Melanoma Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness Exertional (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Temporal Lobe Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major Depression (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Female Genital Tract Fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Period (N=498) | Maintenance Period: Treat to Target (N=219) | Maintenance Period: Routine Care (N=221) | Extension Period: Treat to Target (N=147) | Extension Period: Routine Care (N=176)
Anaemia (Blood and lymphatic system disorders) | 14 (14) | 8 (10) | 11 (13) | 8 (10) | 8 (10)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 3 (3) | 2 (2) | 3 (3) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Dry Eye (Eye disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 4 (5)
Abdominal Distension (Gastrointestinal disorders) | 5 (5) | 3 (4) | 6 (7) | 3 (5) | 6 (8)
Abdominal Pain (Gastrointestinal disorders) | 18 (26) | 23 (31) | 17 (22) | 23 (36) | 22 (34)
Abdominal Pain Upper (Gastrointestinal disorders) | 6 (7) | 7 (7) | 4 (6) | 7 (8) | 4 (8)
Anal Fissure (Gastrointestinal disorders) | 3 (3) | 1 (1) | 6 (6) | 1 (1) | 4 (5)
Anal Fistula (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (5) | 3 (4) | 3 (4)
Constipation (Gastrointestinal disorders) | 7 (8) | 4 (5) | 6 (7) | 4 (5) | 6 (7)
Crohn's Disease (Gastrointestinal disorders) | 9 (10) | 16 (17) | 21 (24) | 18 (19) | 20 (22)
Diarrhoea (Gastrointestinal disorders) | 9 (10) | 11 (13) | 13 (15) | 17 (21) | 17 (24)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (7) | 1 (1) | 5 (9)
Flatulence (Gastrointestinal disorders) | 0 (0) | 4 (5) | 2 (2) | 4 (6) | 4 (4)
Frequent Bowel Movements (Gastrointestinal disorders) | 3 (3) | 2 (2) | 3 (3) | 1 (1) | 5 (5)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 (2) | 4 (4) | 2 (2) | 3 (3) | 4 (4)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (3) | 4 (4)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 6 (8)
Nausea (Gastrointestinal disorders) | 12 (16) | 12 (18) | 12 (15) | 11 (13) | 16 (21)
Toothache (Gastrointestinal disorders) | 3 (3) | 5 (6) | 4 (5) | 6 (7) | 4 (4)
Vomiting (Gastrointestinal disorders) | 7 (10) | 9 (10) | 9 (12) | 5 (6) | 11 (12)
Asthenia (General disorders) | 10 (10) | 8 (8) | 6 (6) | 10 (12) | 8 (8)
Fatigue (General disorders) | 3 (3) | 2 (2) | 7 (8) | 1 (1) | 5 (6)
Influenza Like Illness (General disorders) | 1 (1) | 1 (1) | 0 (0) | 4 (7) | 2 (2)
Pyrexia (General disorders) | 25 (33) | 25 (37) | 19 (21) | 15 (25) | 26 (35)
Anal Abscess (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 5 (5)
Bronchitis (Infections and infestations) | 5 (5) | 4 (7) | 8 (10) | 4 (7) | 11 (15)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 3 (3)
Gastroenteritis (Infections and infestations) | 5 (5) | 7 (7) | 5 (5) | 12 (12) | 9 (9)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 4 (4) | 3 (3) | 3 (3) | 5 (5)
Gastrointestinal Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Influenza (Infections and infestations) | 13 (13) | 12 (13) | 11 (12) | 14 (15) | 14 (16)
Nasopharyngitis (Infections and infestations) | 44 (48) | 29 (48) | 29 (39) | 23 (46) | 35 (58)
Oral Herpes (Infections and infestations) | 6 (6) | 5 (5) | 2 (3) | 4 (6) | 2 (5)
Pharyngitis (Infections and infestations) | 3 (3) | 9 (11) | 7 (7) | 7 (9) | 10 (10)
Rhinitis (Infections and infestations) | 2 (2) | 3 (3) | 4 (5) | 1 (1) | 6 (7)
Sinusitis (Infections and infestations) | 5 (5) | 3 (4) | 2 (2) | 1 (1) | 5 (8)
Tonsillitis (Infections and infestations) | 2 (2) | 3 (3) | 2 (2) | 5 (7) | 4 (5)
Tooth Abscess (Infections and infestations) | 1 (1) | 3 (4) | 2 (3) | 6 (7) | 4 (7)
Upper Respiratory Tract Infection (Infections and infestations) | 6 (7) | 4 (6) | 4 (4) | 4 (6) | 8 (8)
Urinary Tract Infection (Infections and infestations) | 5 (5) | 3 (3) | 4 (7) | 5 (5) | 5 (12)
Vaginal Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 2 (2)
Ligament Sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 4 (4)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 4 (4)
C-Reactive Protein Increased (Investigations) | 6 (6) | 4 (4) | 2 (2) | 3 (3) | 1 (2)
Serum Ferritin Decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 5 (6) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 4 (4) | 4 (4) | 2 (2) | 2 (2) | 4 (4)
Folate Deficiency (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 5 (5) | 4 (4) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 1 (1) | 3 (4) | 1 (1)
Iron Deficiency (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 3 (3) | 3 (3) | 2 (2)
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 2 (2) | 6 (6) | 4 (4)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 2 (2) | 3 (5) | 6 (6) | 6 (9) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 (31) | 24 (30) | 19 (22) | 24 (29) | 26 (35)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 0 (0) | 3 (3) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 7 (8) | 12 (12) | 15 (17) | 18 (25)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 5 (7) | 2 (2) | 6 (8) | 4 (5)
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 4 (4) | 2 (2) | 7 (13)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 36 (47) | 24 (42) | 21 (51) | 20 (62) | 28 (92)
Migraine (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 6 (6)
Anxiety (Psychiatric disorders) | 2 (2) | 4 (4) | 3 (3) | 2 (2) | 6 (6)
Depression (Psychiatric disorders) | 3 (3) | 0 (0) | 5 (5) | 1 (1) | 4 (4)
Insomnia (Psychiatric disorders) | 1 (1) | 4 (4) | 3 (3) | 4 (6) | 5 (5)
Renal Colic (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2) | 3 (4) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 4 (4) | 3 (3) | 2 (2) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (9) | 7 (8) | 6 (8) | 12 (15)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (8) | 5 (5) | 8 (11) | 9 (9)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6) | 5 (5) | 4 (4) | 4 (4) | 4 (4)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 1 (1) | 4 (5) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 4 (5) | 4 (4) | 3 (4) | 4 (6) | 4 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4) | 2 (3) | 5 (5) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (6) | 7 (8) | 9 (10) | 7 (9)
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 1 (1) | 4 (4) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/93/NCT03107793/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/93/NCT03107793/SAP_001.pdf